CLINICAL TRIAL: NCT02972866
Title: Phase III, Multicenter, Randomized, Simple-blinded, Paralel Groups to Evaluate Non Inferiority of Noex® 32µg Versus Budecort Aqua® 32µg in Treatment of Alergic Persistent Rhinitis Moderate to Severe
Brief Title: Clinical Study, Non Inferiority Between Noex® 32µg Versus Budecort Aqua® 32µg in Treatment of Alergic Rhinitis
Acronym: RINEX32
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Regulatory strategy
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EF148
Record Dates: First submitted 2016-11-11; First posted 2016-11-25 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2018-10

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Budesonide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noex 32mcg (Experimental): Noex/Budesonide 32mcg, 2 atomizations in each nostril by the morning and during the night, total of 256 mcg per day.
  Tretament of 28 days.
  Interventions: Drug: Budesonide
- Budecort Aqua 32 mcg (Experimental): Budecort Aqua/Budesonide 32mcg, 2 atomizations in each nostril by the morning and during the night, total of 256 mcg per day.
  Tretament of 28 days.
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — Suspention to nasal use, 2 atomization in each nostril during the morning and at night.
  Other Names: Noex 32mcg; Budecort Aqua 32mcg

SUMMARY:
This study is to evaluate non inferiority of Eurofarma budesonide nasal spary x referral Astrazeneca budesonide. Half patients will receive Eurofarma medication and half patients will receive Astrazeneca medication. There is no placebo group.

DETAILED DESCRIPTION:
Budesonide is a medicine already very used and registered about 20 years. Eurofarma has the intention to collect more data about safety and efficacy and present them to local authority.

This study was draw to treat patients with persisntent rhinits moderate to severe in sites localted locally in Brasil.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 12.
2. History of alergic persistent rhinitis moderate to severe at least 2 years.
3. Proved alergic using PRICK or RAST test.
4. Nasal symptoms (NIS) > 3 and nasal obstruction >1.
5. Indication of nasal corticorteroids use..
6. Washout of nasal corticorteroids for 14 days.
7. ICF.

Exclusion Criteria:

1. Other types of rhinitis;
2. Asthma non controled
3. Use of oral/injectable corticoids 30 days before screening.
4. patients not eligible to complete diaries.
5. patients with alergy to any substance of medicines.
6. non controlled desease.

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Demonstrate non inferiority of Noex comparable with referral product Budecort Aqua in the treatment of rinithis moderate to severe during 4 weeks of treatment. | 28 days
  The questionnaire Nasal Index Score (NIS) will be used to check intensity of symptons and patient will answer this questionnaire daily at home.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Acir Crippa Junior, Principal Investigator — Allergisa Pesquisa Dermato-Cosmética Ltda
Locations (1):
- Allergisa pesquisa dermato-cosmética ltda, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Undecided, but could be shared upon investigator's request.